CLINICAL TRIAL: NCT06286176
Title: Enhancing Breastfeeding Promotion in Lebanon Through a Salutogenic Intervention: A Clinical Trial
Brief Title: Breastfeeding Promotion in Lebanon Through a Salutogenic Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nabiha Ramadan (Other)
Collaborators: Universitat de Girona (Other)
Responsible Party: Sponsor-Investigator, Nabiha Ramadan, M.Sc, Lecturer in Nutrition and Dietetics, Lebanese International University
Organization: Lebanese International University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LIUIRB-200311-NR1
Record Dates: First submitted 2024-02-16; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Breast Feeding; Exclusive Breastfeeding; Salutogenesis
Keywords: Breastfeeding; Salutogenesis; Sense of coherence
MeSH Terms: conditions — Breast Feeding | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: videos (Experimental): 4 videos are created and distributed to subjects in the intervention group. Video 1: 10 days before delivery Video 2: the day of the delivery Video 3: 1 week postpartum Video 4: 1 month postpartum Videos content: encouraging message, information related to breastfeeding management This is arm in applied in all subjects on the intervention group
  Interventions: Behavioral: Videos with breastfeeding education material and encouraging messages
- Behavioral: Whatsapp group (Experimental): 4 Whatsapp groups were created. Each Whatsapp group was moderated by 1 infant feeding helper. Each whatsapp group consisted of 10-15 subjects.
  Mothers asked breastfeeding related questions to infant feeding helpers and also exchange experience with the other mothers on the group.
  This is arm in applied in all subjects on the intervention group. Mothers of the intervention group joined their corresponding whatsapp group 10 days before expected delivery date and the duration of the intervention involving the whatsapp group was until 6 months postpartum.
  Interventions: Behavioral: Whatsapp group

INTERVENTIONS:
Behavioral: Videos with breastfeeding education material and encouraging messages — Distributed videos aim to increase breastfeeding related knowledge and to receive support
  Arms: Behavioral: videos
Behavioral: Whatsapp group — The Whatsapp group is used in the intervention as a platform for interpersonal exchange of information and experience, in addition to peer support.
  Arms: Behavioral: Whatsapp group

SUMMARY:
The study is a randomized control trial to assess the effect of a salutogenic intervention on breastfeeding initiation and duration of exclusive breastfeeding in Lebanon. In this Salutogenic intervention, infant feeding helpers will provide subjects of the intervention group breastfeeding related information , and will support these subjects by counseling and guiding them to find general resistance resources. This aims to increase sense of coherence and its parameters: comprehensibility, manageability and meaningfulness, which are the base of salutogenesis.

DETAILED DESCRIPTION:
Pregnant women were recruited in their 3rd trimester of pregnancy and were randomly assigned to either an intervention or control group.

Both groups received standard breastfeeding education at the maternity ward. Additionally, the intervention is based on informative and supportive videos and a whatsapp group for interpersonal support. Videos and whatsapp groups were created and moderated by Infant Feeding Helpers. These are women from the same socio-economical background as the subjects, and have previous history of breastfeeding a minimum of 6 months exclusive breastfeeding.

The aim of the intervention was to increase initiation and duration of breastfeeding by increasing comprehensibility, manageability and meaningfulness of the breastfeeding period and therefore by enhancing their sense of coherence.

Chi-squared tests were used for descriptive statistics, Wilcoxon test was used for pre- post results of SOC and (SE) within each group. The change in pre-post SOC, SOC parameters and SE scores between control and intervention groups was analyzed with Quade non parametric.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Singleton
* Healthy
* New born not admitted to Neonatal Intensive Care Unit
* Residing in Lebanon

Exclusion Criteria:

* Pregnant with more than 1 fetus
* Mothers with a health condition contraindicating breastfeeding
* Newborn admitted to NICU

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women and breastfeeding mothers
Enrollment: 101 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
breastfeeding initiation | 1 hour after birth
  Number of women who breastfed their infants within 1 hour after birth
Duration of Exclusive breastfeeding | at 6 months postpartum
  number of women who are exclusively breastfeeding at 6 months postpartum. Exclusive breastfeeding indicates feeding infants only breastmilk without any other complementary food nor beverage.

SECONDARY OUTCOMES:
Mean change in Self- esteem in participants from baseline to 6 months postpartum | The first measurement was taken 10 days before delivery and the second measurement was taken at 6 months postpartum
  Measuring the scores of the Rosenberg Self Esteem Scale- 10 items. Scores are from 0 to 30. Higher scores indicate higher self esteem
The Change in Sense of Coherence (SOC) scores from baseline to 6 months postpartum | 1st measurement: 10 days before delivery. 2nd measurement: 6 months postpartum. Score measurements were taken twice per subject for comparison at the end of the intervention.
  The score of the "Sense of Coherence- 13 items" questionnaire. The minimum score is 13, and the maximum score is 91. Higher score indicates higher sense of coherence

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanese International University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Informed consent form, scores of self esteem and scores of sense of coherence
Supporting Information: SAP, ICF, CSR